CLINICAL TRIAL: NCT01665963
Title: Efficacy of TopClosure(C)System in Healing Complicated Pacemaker Wounds
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0042-12-HYMC
Record Dates: First submitted 2012-08-14; First posted 2012-08-16 (Estimated); Last update posted 2012-08-16 (Estimated); Status verified 2012-08

CONDITIONS: Wounds and Injuries
MeSH Terms: conditions — Wounds and Injuries | interventions — Drug Delivery Systems

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TopClosure(c) Treated Wound (Active Comparator): Pressure Bandage using the TopClosure(C) System
  Interventions: Device: TopClosure(c) System
- Traditional Wound Closure Treatment (Active Comparator): Pressure Bandage
  Interventions: Device: Pressure Bandage

INTERVENTIONS:
Device: TopClosure(c) System
  Arms: TopClosure(c) Treated Wound
Device: Pressure Bandage
  Arms: Traditional Wound Closure Treatment

SUMMARY:
Patients receiving oral anticoagulation or anti-platelet therapy are at high risk of hematoma after device implantation. This study intends to examine the efficacy of the TopClosure(c) System in wound healing in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with anticoagulant therapy
* Patients treated with antiplatelet therapy

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Efficacy of TopClosure(c) System | 10 days
  Outside surgeon (blinded) will determine whether wound has healed

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel